CLINICAL TRIAL: NCT00442949
Title: Angioplasty to Blunt the Rise of Troponin in Acute Coronary Syndromes Randomized for an Immediate or Delayed Intervention (The ABOARD Study)
Brief Title: Angioplasty to Blunt the Rise of Troponin in Acute Coronary Syndrome (ACS)
Acronym: ABOARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Myriem CARRIER, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P050705
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2008-04

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; Angioplasty; Abciximab; Troponin release
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Catheterization immediate PCI
  Interventions: Procedure: Catheterization immediate PCI
- 1 (Experimental): delayed PCI
  Interventions: Procedure: delayed PCI

INTERVENTIONS:
Procedure: Catheterization immediate PCI — Catheterization immediate PCI
  Arms: 2
Procedure: delayed PCI — delayed PCI
  Arms: 1

SUMMARY:
Release of troponin evaluated by the peak of troponin during the hospital phase.Because of its sensitivity and specificity as well as its widespread use in routine practice, rise in troponin levels is the main assessment criteria of this study. We plan to demonstrate a significantly altered distribution of the troponin release as evaluated by the peak of troponin for each patient during the hospitalization period (from randomization to cardiologic unit discharge), in the two arms of the trial.

DETAILED DESCRIPTION:
We propose to evaluate the optimal moment for catheterization in patients presenting with acute coronary syndromes by comparing rapid catheterization on the day of admission (within 8 hours of admission, with an average time close to 3 hours, as in the rapid strategy arm of the ISAR-COOL trial) with a slower approach where the examination is scheduled for the next working day (8 to 60 hours post admission, with an average close to 24 hours). Patients included will present with severe unstable angina defined as a TIMI score > 3 All patients must present with an indication for catheterization and they will receive the same optimal pharmacological treatment including abciximab (ReoPro*) when undergoing PCI and started just before the procedure as indicated in the label of the drug (substitution by another drug of the class, eptifibatide or tirofiban, is not possible in the catheterization laboratory according to the labels of these two other drugs). Randomization will evaluate only time to catheterization: rapidly, as soon as possible following admission (within 8 hours of admission) versus a delayed approach (8 to 60 hours following admission). The goal of randomization is to determine the ideal time to catheterization while indications for catheterization, pharmacological treatment, and patient care remain constant. This is a pragmatic study aiming to compare 2 different strategies in the management of ACS.

ELIGIBILITY:
Inclusion Criteria:

1. Man over 18 or non-pregnant woman over 18.
2. Patient hospitalized for severe acute coronary syndrome. To be selected patients will need to have at least 2 criteria for acute coronary syndrome AND a TIMI score > 3 for severity of ACS.

   ACS is defined by at least two of the following diagnostic criteria :
   * ischemic symptom
   * electrocardiographic abnormalities in the ST segment (depression or transitory elevation of at least 0.1 mV), or in the T waves, at least in two contiguous leads positive troponin (as defined locally).

   Severity of ACS is defined by a TIMI score > 3
3. indication for catheterization agreed and possible within the following 8 hours.
4. signed consent form

Exclusion Criteria:

1. Patients that would require immediate catheterization for ongoing refractory ischemia, major arrhythmias, or hemodynamic instability are not eligible for the study.
2. Anticoagulant therapy with antivitamin K within 5 days preceding randomization
3. Thrombolytic therapy during the preceding 24 hours
4. Upstream treatment by a GPIIb/IIIa inhibitor
5. ReoPro should not be administered to patients with known sensitivity to abciximab, to any component of the product or to murine monoclonal antibodies. Because inhibition of platelet aggregation increases the risk of bleeding, ReoPro is contra-indicated in the following clinical situations: active internal bleeding; history of cerebrovascular accident within two years; recent (within two months) intracranial or intraspinal surgery or trauma; recent (within two months) major surgery; intracranial neoplasm, arteriovenous malformation or aneurysm; known bleeding diathesis or severe uncontrolled hypertension; pre-existing thrombocytopenia; vasculitis; hypertensive or diabetic retinopathy; severe hepatic or severe renal failure.
6. Woman nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Release of troponin evaluated by the peak of troponin during the hospital phase | during the hospital phase

SECONDARY OUTCOMES:
Death, MIs and urgent revascularizations will be recorded as ischemic events during 1month following randomization. | during 1month following randomization

CONTACTS AND LOCATIONS:
Overall Officials: Gilles MONTALESCOT, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Institut de Cardiologie - Hôpital Pitié-Salpétrière, Paris, France

REFERENCES:
- [Derived] Barthelemy O, Cayla G, Silvain J, O'Connor SA, Bellemain-Appaix A, Beygui F, Sideris G, Varenne O, Collet JP, Vicaut E, Montalescot G; ABOARD Investigators. Optimal time for catheterization in NSTE-ACS patients with impaired renal function: insights from the ABOARD Study. Int J Cardiol. 2013 Sep 10;167(6):2646-52. doi: 10.1016/j.ijcard.2012.06.126. Epub 2012 Jul 12. PMID 22795712
- [Derived] Montalescot G, Cayla G, Collet JP, Elhadad S, Beygui F, Le Breton H, Choussat R, Leclercq F, Silvain J, Duclos F, Aout M, Dubois-Rande JL, Barthelemy O, Ducrocq G, Bellemain-Appaix A, Payot L, Steg PG, Henry P, Spaulding C, Vicaut E; ABOARD Investigators. Immediate vs delayed intervention for acute coronary syndromes: a randomized clinical trial. JAMA. 2009 Sep 2;302(9):947-54. doi: 10.1001/jama.2009.1267. PMID 19724041